CLINICAL TRIAL: NCT07390487
Title: The Effects of Audio-Based Therapy on Anxiety in Psoriasis
Acronym: PsOUND-PSO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PsOUND-PSO
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis (PsO); Anxiety
Keywords: Surveys and Questionnaires; Acoustic Stimulation; Complementary Therapies
MeSH Terms: conditions — Psoriasis; Anxiety Disorders | interventions — Music Therapy; Complementary Therapies; Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): Participants listen to the iso-principle music with added auditory beat stimulation playlist for 23-30 minutes.
  Interventions: Behavioral: Music Therapy
- Pink Noise (Sham Comparator): Participants listen to the pink noise playlist for 23-30 minutes.
  Interventions: Behavioral: Pink Noise

INTERVENTIONS:
Behavioral: Music Therapy — Participants listen to the iso-principle music with added auditory beat stimulation playlist for 23-30 minutes.
  Other Names: Music therapy and auditory beat stimulation (ABS); Music; Complementary Therapy; Complementary Therapies; Acoustic Stimulation
  Arms: Music Therapy
Behavioral: Pink Noise — Participants listen to the pink noise playlist for 23-30 minutes.
  Arms: Pink Noise

SUMMARY:
Anxiety in psoriasis is associated with impaired quality of life, and the prevalence of anxiety symptoms in psoriatic populations is approximately 34% and anxiety disorders up to 16%. Many experts recommend routine screening, referral, and interventions for anxiety in psoriasis; however, many barriers inhibit access to mental health resources and proper management. To our knowledge, there is a lack of easily accessible interventions that manage anxiety. Audio-based therapy offers convenient and effective interventions that show reduced anxiety in published, randomized studies and is a promising management for psoriasis patients. This study will evaluate the effects of audio therapy in patients with psoriasis and measure changes in overall symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Self-reported dermatologist-diagnosed psoriasis
* GAD 2-Item Score ≥1 at screening
* Ability to consent and complete pre- and post-intervention surveys.
* Internet access and the ability to use a computer/smartphone with headphones for a single 23-30 minute session at home.

Exclusion Criteria:

* Severe hearing impairment precluding headphone listening
* Any condition requiring strict sound avoidance (such as seizure/epilepsy, major head trauma, severe sound-triggered migraine) that would make participation unsafe.
* Other diagnoses that in the investigator's judgment preclude safe participation or interfere with anxiety or psoriasis evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety: State Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | From the pre-intervention survey to the post-intervention survey, approximately 30 minutes.
  The STICSA has good reliability and validity as a measure of state and trait cognitive and somatic anxiety. In this study, the post-intervention anxiety score is subtracted from the pre-intervention anxiety score, giving a measure of anxiety reduction. Greater anxiety reduction scores would indicate a better anxiety outcome.

SECONDARY OUTCOMES:
Mood: Positive and Negative Affect Scale (PANAS) | From the pre-intervention survey to the post-intervention survey, approximately 30 minutes.
  The PANAS has demonstrated good reliability and validity, and has been widely used in numerous studies to assess mood. In this study, the post-intervention PANAS scores are subtracted from the pre-intervention PANAS scores, giving a measure of positive and negative mood changes. The scale generates two scores: 1) Positive affect (higher score indicates better mood outcome) and 2) Negative affect (higher score indicates worse mood outcome).
Itch: Itch Numeric Rating Score (INRS) | From the pre-intervention survey to the post-intervention survey, approximately 30 minutes.
  The INRS has good reliability and validity as a measure of 24-hour itch severity, though validity testing over more acute intervals remains limited. In this study, the post-intervention itch score is subtracted from the pre-intervention itch score, giving a measure of itch reduction. Greater itch reduction scores may indicate a better itch outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Liao, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Liao Lab at UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yan D, Blauvelt A, Dey AK, Golpanian RS, Hwang ST, Mehta NN, Myers B, Shi ZR, Yosipovitch G, Bell S, Liao W. New Frontiers in Psoriatic Disease Research, Part II: Comorbidities and Targeted Therapies. J Invest Dermatol. 2021 Oct;141(10):2328-2337. doi: 10.1016/j.jid.2021.02.743. Epub 2021 Apr 19. PMID 33888321
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Riew GJ, Kamal K, Hijaz B, Awh KC, Nambudiri VE. Clinical music interventions and music therapy in dermatology. Arch Dermatol Res. 2023 Nov;315(9):2485-2490. doi: 10.1007/s00403-023-02634-1. Epub 2023 May 19. PMID 37208459
- [Background] Mallik A, Russo FA. The effects of music & auditory beat stimulation on anxiety: A randomized clinical trial. PLoS One. 2022 Mar 9;17(3):e0259312. doi: 10.1371/journal.pone.0259312. eCollection 2022. PMID 35263341
- [Background] Jalenques I, Bourlot F, Martinez E, Pereira B, D'Incan M, Lauron S, Rondepierre F. Prevalence and Odds of Anxiety Disorders and Anxiety Symptoms in Children and Adults with Psoriasis: Systematic Review and Meta-analysis. Acta Derm Venereol. 2022 Aug 26;102:adv00769. doi: 10.2340/actadv.v102.1386. PMID 35604236
- [Background] Hedemann TL, Liu X, Kang CN, Husain MI. Associations between psoriasis and mental illness: an update for clinicians. Gen Hosp Psychiatry. 2022 Mar-Apr;75:30-37. doi: 10.1016/j.genhosppsych.2022.01.006. Epub 2022 Jan 25. PMID 35101785
- [Background] Gros DF, Antony MM, Simms LJ, McCabe RE. Psychometric properties of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA): comparison to the State-Trait Anxiety Inventory (STAI). Psychol Assess. 2007 Dec;19(4):369-81. doi: 10.1037/1040-3590.19.4.369. PMID 18085930
- [Background] Phan NQ, Blome C, Fritz F, Gerss J, Reich A, Ebata T, Augustin M, Szepietowski JC, Stander S. Assessment of pruritus intensity: prospective study on validity and reliability of the visual analogue scale, numerical rating scale and verbal rating scale in 471 patients with chronic pruritus. Acta Derm Venereol. 2012 Sep;92(5):502-7. doi: 10.2340/00015555-1246. PMID 22170091
- [Background] Gray EK, Watson, D. Assessing positive and negative affect via self-report. In: Coan JA, Allen, J.J.B., editor. Handbook of emotion elicitation and assessment. New York, NY: Oxford University Press; 2007.
- [Background] Bados A, Gomez-Benito J, Balaguer G. The state-trait anxiety inventory, trait version: does it really measure anxiety? J Pers Assess. 2010 Nov;92(6):560-7. doi: 10.1080/00223891.2010.513295. PMID 20954057